CLINICAL TRIAL: NCT01400503
Title: An Open-label, Multicenter Study to Evaluate the Safety of Long-term Treatment With Siltuximab in Subjects With Multicentric Castleman's Disease
Brief Title: A Study to Evaluate the Safety of Long-term Treatment With Siltuximab in Patients With Multicentric Castleman's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018469; CNTO328MCD2002 (Other: Janssen Research & Development, LLC); 2010-022837-27 (EudraCT Number)
Record Dates: First submitted 2011-04-21; First posted 2011-07-22 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Multicentric Castleman's Disease
Keywords: Multicentric Castleman's Disease; Multicentric; Castleman; Siltuximab; Long term safety
MeSH Terms: conditions — Multi-centric Castleman's Disease | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Siltuximab (Experimental): Siltuximab 11 mg/kg, intravenous infusion, given as a 1-hour infusion every 3 weeks.
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Type=exact number, unit=mg/kg, number=11, form=intravenous solution, route=intravenous. Siltuximab given as a 1-hour infusion every 3 weeks.

SUMMARY:
The purpose of this study is to evaluate the long-term safety of siltuximab in patients with multicentric Castleman's disease (MCD).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (study conducted in multiple sites), non-randomized (patients are not assigned by chance to treatment groups), Phase 2b study. Up to 75 patients with MCD will be eligible for the study, the majority of whom will be on active therapy with siltuximab at the time of enrollment. Patients will be either siltuximab-naive or have not progressed on siltuximab in the opinion of the investigator. Duration of disease control and survival will be assessed. Data collection for patients who discontinue treatment will be limited to survival, occurrence of malignancies, and subsequent therapies for MCD, which will be assessed twice per year until the patient has been lost to follow up or has withdrawn consent for the study, whichever occurs first. An interim analysis will be conducted (no later than 2 years after the start of enrollment) to further evaluate the benefit and safety of long-term treatment with siltuximab in patients with MCD. A data will occur at 6 years after the start of enrollment and for those patients remaining on treatment after the data cutoff, data collection will be limited to pregnancies and serious adverse events (SAEs), including information on study agent administration and concomitant medications associated with an SAE. Safety evaluations for adverse events, clinical laboratory tests, vital signs, and physical examination will be performed throughout the study. The end of study is the date of the last assessment for the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Has multicentric Castleman's disease
* Have previously been enrolled in Study C0328T03 or CNTO328MCD2001 (either treatment arm)
* Have had their last administration of study treatment (siltuximab or placebo) less than 6 weeks (window of plus 2 weeks) prior to first dose
* Patients must not have had disease progression while receiving siltuximab. For those patients originally assigned to placebo in the CNTO328MCD2001 study, patients who have received less than 4 months of siltuximab following crossover will also be eligible
* Have adequate clinical laboratory parameters within 2 weeks prior to the first dose of siltuximab for this study

Exclusion Criteria:

* Unmanageable toxicity, an adverse event, progression of disease, or withdrawal of consent as reason for discontinuing treatment from previous sponsor-initiated siltuximab study
* Vaccination with live, attenuated vaccines within 4 weeks of first dose of this study
* Known unmanageable allergies, hypersensitivity, intolerance to monoclonal antibodies, to murine, chimeric, human proteins or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (26):
- United States (7):
  - Little Rock, Arkansas
  - Tampa, Florida
  - Lansing, Michigan
  - Chapel Hill, North Carolina
  - Greenville, South Carolina
  - Houston, Texas
  - Seattle, Washington
- Leuven, Belgium
- São Paulo, Brazil
- Toronto, Canada
- China (2):
  - Beijing
  - Chengdu
- Cairo, Egypt
- France (3):
  - Montpellier
  - Tours
  - Vandœuvre-lès-Nancy
- Berlin, Germany
- Shatin, Hong Kong
- Ramat Gan, Israel
- Auckland, New Zealand
- Oslo, Norway
- Singapore, Singapore
- Seoul, South Korea
- Madrid, Spain
- Taipei, Taiwan
- Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled in this study CNTO328MCD2002 included participants who were previously enrolled in study C0328T03 (NCT00412321) or CNTO328MCD2001 (NCT01024036) (either placebo or siltuximab treatment arm). A total of 60 participants from previous MCD studies C0328T03 and CNTO328MCD2001 were found eligible to be enrolled in this study.
Groups:
- Siltuximab: Participants received siltuximab 11 milligram per kilogram (mg/kg) as a 1-hour intravenous infusion every 3 weeks until disease progression, withdrew, experienced unacceptable toxicity,or until the 6-year data cutoff, whichever occurred first.
Period: Overall Study
Arm/Group | Siltuximab
Started | 60
Completed | 0
Not Completed | 60
Not completed — Withdrawal by Subject | 1
Not completed — Study Terminated by Sponsor | 58
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Siltuximab
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 3
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 23
  Black or African American | 3
  Hispanic or Latino | 5
  Other | 3
  White Non-Hispanic | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1
  Brazil | 1
  Canada | 1
  China | 6
  Egypt | 1
  France | 3
  Germany | 1
  Hong Kong | 3
  New Zealand | 2
  Norway | 2
  Singapore | 3
  Korea, Republic Of | 4
  Spain | 2
  Taiwan, Province Of China | 1
  United Kingdom | 2
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 6 years
Population: Safety analysis set included all enrolled participants in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Siltuximab
Number analyzed (Participants) | 60
Participants | 60

2. Secondary Outcome: Percentage of Previously Responding Participants Who Maintained Disease Control
Description: Percentage of participants maintaining disease control (defined as stable or better response) was defined as the percentage of previously responding participants who had not progressed during the long-term safety extension based on investigator assessment. A worsening in any of the measures will be considered as a progression of the disease.
Time Frame: Up to 6 years
Population: Population included subset of safety analysis set who previously responded to siltuximab treatment ie, did not report disease progression while receiving siltuximab in study C0328T03 or CNTO328MCD2001.
Measure: Number; unit: percentage of participants
Arm/Group | Siltuximab
Number analyzed (Participants) | 57
percentage of participants | 96.5

3. Secondary Outcome: Percentage of Siltuximab-naive Participants Who Experienced Disease Control
Description: Percentage of participants experiencing disease control was defined as the percentage of siltuximab-naïve participants who had stable or better response during the long-term safety extension based on investigator's judgment. Disease control was defined as stable or better response assessed by the investigators.
Time Frame: Up to 6 years
Population: Population included subset of safety analysis set who were previously Siltuximab-naive i.e., received placebo in study CNTO328MCD2001 and never received siltuximab prior to enrollment in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Siltuximab
Number analyzed (Participants) | 3
percentage of participants | 100

4. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control (DODC) was defined as the time from the first siltuximab administration in this study to disease progression as assessed by the investigator. Disease control was defined as stable or better response assessed by the investigators. Kaplan-Meier method was used to estimate the duration of disease control.
Time Frame: Up to 6 years
Population: Safety analysis set included all enrolled participants in this study.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Siltuximab
Number analyzed (Participants) | 60
years | NA [NA to NA] — Median and confidence interval (CI) were not estimable due to insufficient number of participants with loss of response or disease control (due to high censorship rate).

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time between the first study siltuximab administration and death due to any cause. Kaplan-Meier method was used to estimate the overall survival.
Time Frame: Up to 6 years
Population: Safety analysis set included all enrolled participants in this study.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Siltuximab
Number analyzed (Participants) | 60
years | NA [NA to NA] — Median and CI were not estimable due to insufficient number of participants with death.

6. Secondary Outcome: Number of Participants Positive for Antibodies to Siltuximab
Description: Serum samples were screened for antibodies binding to siltuximab and number of participants positive for antibodies to siltuximab was reported.
Time Frame: Up to 6 years
Population: Safety analysis set included all enrolled participants in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Siltuximab
Number analyzed (Participants) | 60
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: Safety analysis set included all enrolled participants in this study.
Arm/Group | Siltuximab
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 25/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=60)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Polycythaemia (Blood and lymphatic system disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Vitreous Haemorrhage (Eye disorders) | 1
Food Poisoning (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Umbilical Hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Abscess Limb (Infections and infestations) | 1
Anal Abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Lower Respiratory Tract Infection (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Vulval Abscess (Infections and infestations) | 1
Wound Infection Staphylococcal (Infections and infestations) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Avulsion Fracture (Injury, poisoning and procedural complications) | 1
Chest Injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fractured Sacrum (Injury, poisoning and procedural complications) | 1
Ilium Fracture (Injury, poisoning and procedural complications) | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 2
Tibia Fracture (Injury, poisoning and procedural complications) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1
Benign Neoplasm of Testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrospinal Fluid Leakage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Bladder Pain (Renal and urinary disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Micturition Disorder (Renal and urinary disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
Ureteral Disorder (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 1
Mastectomy (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Hypertensive Crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=60)
Anaemia (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Atrioventricular Block First Degree (Cardiac disorders) | 2
Cardiac Disorder (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 6
Tinnitus (Ear and labyrinth disorders) | 5
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 6
Cataract (Eye disorders) | 4
Dry Eye (Eye disorders) | 2
Eye Irritation (Eye disorders) | 2
Periorbital Oedema (Eye disorders) | 2
Vision Blurred (Eye disorders) | 7
Abdominal Discomfort (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 14
Abdominal Pain Lower (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 10
Anal Fistula (Gastrointestinal disorders) | 2
Aphthous Ulcer (Gastrointestinal disorders) | 5
Chronic Gastritis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 17
Dental Caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 23
Dry Mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 9
Gingival Pain (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Hiatus Hernia (Gastrointestinal disorders) | 3
Mouth Ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 22
Oral Pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Tongue Ulceration (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 3
Catheter Site Pain (General disorders) | 2
Chest Discomfort (General disorders) | 2
Chest Pain (General disorders) | 3
Cyst (General disorders) | 2
Fatigue (General disorders) | 31
Generalised Oedema (General disorders) | 4
Influenza Like Illness (General disorders) | 2
Localised Oedema (General disorders) | 3
Malaise (General disorders) | 8
Oedema (General disorders) | 2
Oedema Peripheral (General disorders) | 13
Pain (General disorders) | 7
Peripheral Swelling (General disorders) | 5
Pyrexia (General disorders) | 6
Cholelithiasis (Hepatobiliary disorders) | 2
Gallbladder Polyp (Hepatobiliary disorders) | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 11
Hyperbilirubinaemia (Hepatobiliary disorders) | 7
Seasonal Allergy (Immune system disorders) | 5
Acute Sinusitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 4
Ear Infection (Infections and infestations) | 6
Fungal Infection (Infections and infestations) | 3
Furuncle (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 8
Herpes Simplex (Infections and infestations) | 2
Herpes Zoster (Infections and infestations) | 5
Influenza (Infections and infestations) | 6
Laryngitis (Infections and infestations) | 3
Localised Infection (Infections and infestations) | 2
Lower Respiratory Tract Infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 11
Onychomycosis (Infections and infestations) | 2
Oral Candidiasis (Infections and infestations) | 2
Oral Herpes (Infections and infestations) | 2
Otitis Media (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 4
Rash Pustular (Infections and infestations) | 5
Respiratory Tract Infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 10
Skin Infection (Infections and infestations) | 3
Tinea Infection (Infections and infestations) | 2
Tooth Abscess (Infections and infestations) | 3
Tooth Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 40
Urinary Tract Infection (Infections and infestations) | 11
Viral Infection (Infections and infestations) | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 5
Hand Fracture (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 5
Procedural Pain (Injury, poisoning and procedural complications) | 4
Skin Abrasion (Injury, poisoning and procedural complications) | 5
Tibia Fracture (Injury, poisoning and procedural complications) | 2
Tooth Fracture (Injury, poisoning and procedural complications) | 3
Alanine Aminotransferase Increased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 4
Blood Creatinine Increased (Investigations) | 4
Blood Fibrinogen Decreased (Investigations) | 3
Blood Phosphorus Increased (Investigations) | 2
Haemoglobin Increased (Investigations) | 4
Protein Total Decreased (Investigations) | 3
Serum Ferritin Decreased (Investigations) | 4
Weight Decreased (Investigations) | 4
Weight Increased (Investigations) | 11
Decreased Appetite (Metabolism and nutrition disorders) | 13
Enzyme Abnormality (Metabolism and nutrition disorders) | 5
Gout (Metabolism and nutrition disorders) | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 17
Hyperuricaemia (Metabolism and nutrition disorders) | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 20
Back Pain (Musculoskeletal and connective tissue disorders) | 19
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 3
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 14
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 2
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 2
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Amnesia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 14
Hypoaesthesia (Nervous system disorders) | 5
Memory Impairment (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 6
Peripheral Motor Neuropathy (Nervous system disorders) | 5
Peripheral Sensory Neuropathy (Nervous system disorders) | 15
Polyneuropathy (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 11
Nightmare (Psychiatric disorders) | 2
Azotaemia (Renal and urinary disorders) | 4
Dysuria (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 3
Renal Impairment (Renal and urinary disorders) | 6
Urinary Retention (Renal and urinary disorders) | 2
Erectile Dysfunction (Reproductive system and breast disorders) | 3
Menorrhagia (Reproductive system and breast disorders) | 2
Pelvic Pain (Reproductive system and breast disorders) | 3
Prostatitis (Reproductive system and breast disorders) | 2
Prostatomegaly (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 15
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 3
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Eczema (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9
Night Sweats (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 19
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 21
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 16
Rash Pruritic (Skin and subcutaneous tissue disorders) | 3
Scar Pain (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Skin Induration (Skin and subcutaneous tissue disorders) | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4
Vitiligo (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 7
Hot Flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 15
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2014-04-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT01400503/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT01400503/SAP_001.pdf